CLINICAL TRIAL: NCT00338286
Title: A Randomized, Open-label, Multicenter, Phase 3 Study of Epoetin Alfa Plus Standard Supportive Care Versus Standard Supportive Care in Anemic Patients With Metastatic Breast Cancer Receiving Standard Chemotherapy
Brief Title: A Study of Epoetin Alfa Plus Standard Supportive Care Versus Standard Supportive Care Only in Anemic Patients With Metastatic Breast Cancer Receiving Standard Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR005143; EPOANE3010 (Other: Janssen Research & Development, LLC); CR005143 (Other: Janssen Research & Development, LLC); 2005-001817-17 (EudraCT Number: Janssen Research & Development, LLC)
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Results first posted 2016-03-24 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2018-02

CONDITIONS: Breast Cancer; Neoplasm Metastasis
Keywords: anemia; metastatic breast cancer; Hemoglobin; progression-free survival (PFS); erythropoiesis-stimulating agents (ESA)
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Anemia | interventions — Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- 001 (Experimental): epoetin alfa + packed RBC transfusion 40 000 IU SC once a week.
  Interventions: Drug: epoetin alfa + packed RBC transfusion
- 002 (Other): Standard supportive care (packed RBC transfusion) Per doctor prescription
  Interventions: Other: Standard supportive care (packed RBC transfusion)

INTERVENTIONS:
Other: Standard supportive care (packed RBC transfusion) — Per doctor prescription
  Arms: 002
Drug: epoetin alfa + packed RBC transfusion — 40,000 IU SC once a week.
  Arms: 001

SUMMARY:
The purpose of this study is to assess the impact on tumor progression as evaluated by progression-free survival (PFS) of epoetin alfa plus standard supportive care as compared with standard supportive care alone (packed red blood cell (RBC) transfusions), for treating anemia according to label guidance in patients with metastatic breast cancer receiving standard chemotherapy.

DETAILED DESCRIPTION:
Anemia is a common complication of the treatment of metastatic breast cancer and is related to the effects of chemotherapy and to chronic disease itself. This is a randomized, open-label, multicenter, international study to further examine the safety of the study drug used with standard supportive care (i.e., packed RBC transfusions) compared to standard supportive care alone, when used to treat anemia associated with chemotherapy. This study will be done in subjects with metastatic breast cancer who are being or will be treated with first-line chemotherapy with standard dose schedules of taxane monotherapy, or a taxane plus trastuzumab, or an anthracycline plus either a taxane or cyclophosphamide. The study hypothesis is that epoetin alfa, when used as supportive anemia care, does not increase the risk of tumor progression or death. The study treatment will be compared to the control treatment by comparing progression-free survival, i.e., the number of months from the date a patient is randomized into the trial to the date of the first documented disease progression or death. In addition to their chemotherapy, half of the subjects will be assigned to receive study drug (epoetin alfa) and half of the subjects will be assigned to standard supportive care for anemia. Subjects treated with the study drug will receive standard supportive care (packed RBC transfusions) plus 40,000 IU epoetin alfa given subcutaneously once a week until 4 weeks after the last cycle of chemotherapy or until disease progression, whichever comes first.The hypothesis is to test that epoetin alfa, when used as supportive anemia care, is non-inferior to control (standard supportive care alone), as measured by progression free survival (PFS). Patients treated with the study drug will receive standard supportive care (packed red blood cells (RBC) transfusions) plus 40,000 IU epoetin alfa given subcutaneously once a week until 4 weeks after the last cycle of chemotherapy or until disease progression, whichever comes first. Dose adjustments (dose escalation, dose reduction, dose interruption, and dose resumption) of epoetin alfa will be based on hemoglobin (Hb) and confirm to prescribing information.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed (e.g., slide of tissue) breast cancer
* HER2/NEU positive or negative
* Clinical evidence of metastasis (e.g., biopsy) with at least 1 measurable metastatic (M1) lesion prior to starting the current chemotherapy
* Received 1st and 2nd line chemotherapy
* Hemoglobin (Hb) <= 11g/dL at the time of randomization
* planned to receive at least 2 more cycles of chemotherapy
* Life expectancy > 6 months
* Eastern Cooperative Oncology Group score 0 or 1
* At least 18 years old using effective birth control or surgically sterile or postmenopausal for 1 year

Exclusion Criteria:

* Active second cancer
* no recent history of clinically relevant thrombovascular event
* Current treatment with anticoagulants
* Brain metastasis or CNS involvement
* Anemia secondary to another cause
* Recent (within prior 1 months) use of an ESA
* Patient pregnant or breast feeding
* Progressive disease during adjuvant/neoadjuvant chemotherapy
* Rapidly progressive or life-threatening metastatic disease
* Concomitant endocrine therapy
* Patient in whom the only site of metastasis was local and was successfully treated surgically.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2098 (Actual)
Dates: Start 2006-03-02 (Actual); Primary Completion 2014-07-07 (Actual); Study Completion 2017-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC C. Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (174):
- United States (14):
  - Anaheim, California
  - Gainesville, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - Rockledge, Florida
  - Hazard, Kentucky
  - Alexandria, Louisiana
  - Marrero, Louisiana
  - Jackson, Mississippi
  - Lake Success, New York
  - Staten Island, New York
  - Philadelphia, Pennsylvania
  - Corpus Christi, Texas
  - Houston, Texas
- Argentina (9):
  - Buenos Aires
  - Capital Federal
  - Ciudad Autonoma de Buenos Airess
  - Córdoba
  - La Plata
  - Mendoza
  - Quilmes
  - Rosario
  - Santa Fe
- Brazil (12):
  - Barretos
  - Curitiba
  - Goiânia/Go
  - Ijuí
  - Jaú
  - Piracicaba
  - Porto Alegre
  - Ribeirão Preto/Sp
  - Santo André
  - São José do Rio Preto
  - São Paulo
  - São Paulol
- Bulgaria (5):
  - Plovdiv
  - Rousse
  - Sofia
  - Stara Zagora
  - Varna
- Chile (5):
  - Arica
  - Santiago
  - Temuco
  - Valdivia
  - Valparaíso
- Colombia (3):
  - Bogotá
  - Floridablanca-Santander
  - Montería
- Ecuador (4):
  - Cuenca
  - Guayaquil
  - Portoviejo
  - Quito
- Georgia (2):
  - Batumi
  - Tbilisi
- New Territories, Hong Kong
- India (22):
  - Ahmedabad
  - Andra Pradesh
  - Bangalore
  - Bengaluru
  - Bhopal
  - Delhi
  - Hyderabad
  - Jaipur
  - Kārnād
  - Kerala
  - Kochi
  - Kolkata
  - Mangalore
  - Mumbai
  - Nashik
  - New Delhi
  - Pune
  - Tamil Nadu Na
  - Tamil Nadu
  - Thiruvananthapuram
  - Uttar Pradesh
  - Vellore
- Indonesia (4):
  - Bandung
  - Jakarta
  - Semarang
  - Yogyakarta
- Malaysia (5):
  - George Town
  - Kampung Baharu Nilai
  - Kelantan
  - Kuala Lumpur
  - Tanjung Bungah
- Mexico (9):
  - Chihuahua City
  - Guerrero
  - León
  - Mérida
  - Morelia
  - Puebla City
  - San Luis Potosí City
  - Sinaloa
  - Zapopan
- North Macedonia (2):
  - Bitola
  - Skopje
- Philippines (5):
  - Cebu
  - Davao City
  - Iloilo City
  - Manila
  - Quezon City
- Poland (9):
  - Bialystok
  - Gdansk
  - Gliwice
  - Katowice
  - Krakow
  - Lodz
  - Olsztyn
  - Poznan
  - Wroclaw
- Romania (8):
  - Brasov
  - Bucharest
  - Cluj-Napoca
  - Iași
  - Onești
  - Sibiu
  - Suceava
  - Timișoara
- Russia (24):
  - Arkhangelsk
  - Balashikha
  - Belgorod
  - Chelyabinsk
  - Engels Saratov Region
  - Ivanovo
  - Kazan'
  - Krasnodar
  - Leningrad Region
  - Lipetsk
  - Magnitogorsk
  - Moscow
  - Novosibirsk
  - Obninsk
  - Orenburg
  - Perm
  - Pyatigorsk
  - Ryazan
  - Saint Petersburg
  - Smolensk
  - Tyumen
  - Ufa
  - Voronezh
  - Yekaterinburg
- South Africa (7):
  - Bloemfontein
  - Cape Town
  - Durban
  - Johannesburg
  - Klerksdorp
  - Port Elizabeth
  - Pretoria
- Taiwan (8):
  - Changhua
  - Chiayi City
  - Hualien City
  - Kaohsiung City
  - Taichung
  - Tainan
  - Taipei
  - Taoyuan District
- Ukraine (16):
  - Cherkassy
  - Chernihiv
  - Chernivtsi
  - Dnipro
  - Donetsk
  - Ivano-Francovsk
  - Kharkiv
  - Kiev
  - Lviv
  - Odesa
  - Poltava
  - Sumy
  - Uzhhorod
  - Vinnitsa
  - Vinnytsia
  - Zaporizhzhya

REFERENCES:
- [Derived] Leyland-Jones B, Bondarenko I, Nemsadze G, Smirnov V, Litvin I, Kokhreidze I, Abshilava L, Janjalia M, Li R, Lakshmaiah KC, Samkharadze B, Tarasova O, Mohapatra RK, Sparyk Y, Polenkov S, Vladimirov V, Xiu L, Zhu E, Kimelblatt B, Deprince K, Safonov I, Bowers P, Vercammen E. A Randomized, Open-Label, Multicenter, Phase III Study of Epoetin Alfa Versus Best Standard of Care in Anemic Patients With Metastatic Breast Cancer Receiving Standard Chemotherapy. J Clin Oncol. 2016 Apr 10;34(11):1197-207. doi: 10.1200/JCO.2015.63.5649. Epub 2016 Feb 8. PMID 26858335

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants in safety data were grouped as treatment actually received (3 were assigned to SOC but received epoetin alfa; 2 were assigned to EPO, but received SOC) so, 1 more to EPO (1051) 1 less in SOC (1045) actually received treatment. Efficacy, safety were analyzed by 1050 (EPO), 1048 (SOC), 1051 (EPO), 1045 (SOC) respectively.
Groups:
- Standard Supportive Care (SOC): Participants received standard supportive care as packed red blood cells (RBC) transfusion as per Investigator's discretion
- Epoetin Alfa: Participants received SOC plus epoetin alfa 40,000 international units (IU) subcutaneously (SC) once a week.
Period: Overall Study
Arm/Group | Standard Supportive Care (SOC) | Epoetin Alfa
Started | 1048 | 1050
Completed | 815 | 837
Not Completed | 233 | 213
Not completed — Withdrawal by Subject | 50 | 54
Not completed — Lost to Follow-up | 80 | 66
Not completed — Other | 103 | 93

BASELINE CHARACTERISTICS:
Population: The intent to treat (ITT) population included all participants who were randomized in either Standard of Care (SOC) or Epoetin alfa group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Supportive Care (SOC) | Epoetin Alfa | Total
Number analyzed (Participants) | 1048 | 1050 | 2098
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (10.54) | 51.9 (10.49) | 51.9 (10.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1048 | 1050 | 2098
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 4 | 5 | 9
  BRAZIL | 27 | 16 | 43
  BULGARIA | 14 | 10 | 24
  CHILE | 11 | 13 | 24
  COLOMBIA | 3 | 1 | 4
  ECUADOR | 1 | 1 | 2
  GEORGIA | 241 | 200 | 441
  HONG KONG | 1 | 0 | 1
  INDIA | 211 | 237 | 448
  INDONESIA | 4 | 5 | 9
  MACEDONIA | 4 | 5 | 9
  MALAYSIA | 7 | 6 | 13
  MEXICO | 8 | 12 | 20
  PHILIPPINES | 60 | 54 | 114
  ROMANIA | 0 | 3 | 3
  RUSSIA | 102 | 129 | 231
  TAIWAN | 19 | 30 | 49
  UKRAINE | 328 | 318 | 646
  UNITED STATES OF AMERICA | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression free survival was based in investigator-determined progressive disease (PD) and calculated from the date of randomization to the date of PD or the date of death, whichever occurred first. Participants who had not progressed and were still alive at the time of clinical cut off were censored at the last disease assessment prior to the clinical cutoff. For PD or death with a missing interval immediately preceding the event, progression-free survival (PFS) was censored at the last disease assessment prior to the missing interval. Participants who withdrew from the study (withdrawal of consent or lost to follow-up) without progression were censored at the time of the last disease assessment.
Time Frame: From the date of randomization to the date of disease progression (PD) or death, whichever occurred first (up to 8.4 years)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Standard of Care (SOC): Participants received standard supportive care as packed red blood cells (RBC) transfusion as per Investigator's discretion.
Arm/Group | Standard of Care (SOC) | Epoetin Alfa
Number analyzed (Participants) | 1048 | 1050
Months | 7.4 [7.1 to 7.6] | 7.4 [6.9 to 7.6]

2. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was defined as the interval between the date of randomization to the date of death from any cause. For participants who were lost to follow-up or withdrew before the final database lock, OS was censored at the last date the participants was known to be alive. For participants who were still alive and on study at the time of the final database lock, OS was censored at the date of final database lock.
Time Frame: From randomization up to death from any cause (up to 8.4 years)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Standard of Care (SOC) | Epoetin Alfa
Number analyzed (Participants) | 1048 | 1050
Months | 18.0 [16.6 to 19.6] | 17.8 [16.6 to 19.1]

3. Secondary Outcome: Time to Tumor Progression
Description: The Time to tumor progression (TTP) was defined as the time from the date of starting treatment until the date of first documented evidence of progression of tumor. TTP was measured from the date of randomization to the date of the first documented PD (including death due to PD without prior PD).
Time Frame: From date of randomization to the date of the first documented PD (up to 8.4 years)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Standard of Care (SOC) | Epoetin Alfa
Number analyzed (Participants) | 1048 | 1050
Months | 7.5 [7.4 to 8.0] | 7.5 [7.4 to 7.9]

4. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall response was RECIST criteria. Complete response (CR) is appearance of all target and non-target lesions. Partial response (PR):a) 30% decrease in sum of lactate dehydrogenase(LD) of target lesions from baseline OR b) complete disappearance of target lesions, with persistence of one or more non-target measurable lesion or one or more non-measurable, evaluable lesions. Progressive disease(PD):a) 20% increase in sum of LDs of target lesions, taking as reference smallest sum LD recorded since treatment started; OR b) appearance of one or more new lesions or a clear worsening of measurable non-target lesions or evaluable disease with stable measurable lesions. Stable disease (SD):a) sufficient shrinkage to qualify for PR;b) sufficient increase to qualify for PD. Non evaluable(NE) lesion: all other lesions, including small lesions (longest diameter <20 millimeter (mm) with conventional techniques or <10 mm with spiral CT scan) and truly non-measurable lesions.
Time Frame: every 8 weeks for 1 year and then every 12 weeks until PD or death, whichever occurred first (up to 8.4 years)
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Standard of Care (SOC) | Epoetin Alfa
Number analyzed (Participants) | 1048 | 1050
Percentage of participants
  Complete response (CR) | 3 | 3
  Partial response (PR) | 48 | 47
  Stable disease (SD) | 30 | 32
  Progressive disease (PD) | 13 | 12
  Not evaluable (NE) | 1 | 2
  Not available (NA) | 5 | 5

5. Secondary Outcome: Percentage of Participants With Suspected Thrombotic Vascular Events (TVEs)
Description: Suspected TVEs were identified by investigators and relevant clinical information was collected.
Time Frame: up to 8.4 years
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Standard of Care (SOC) | Epoetin Alfa
Number analyzed (Participants) | 1048 | 1050
Percentage of participants | 3.72 | 4.86

ADVERSE EVENTS:
Time Frame: From randomization up to 8.4 years
Description: The Safety analysis set included included all randomized participants for whom safety assessment data were available. Participants in the safety population were grouped according to the treatment actually received.
Arm/Group | Standard Supportive Care (SOC) | Epoetin Alfa
Serious Adverse Events (participants affected / at risk) | 229/1045 | 251/1051
Other Adverse Events (participants affected / at risk) | 883/1045 | 898/1051
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Supportive Care (SOC) (N=1045) | Epoetin Alfa (N=1051)
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 15 | 10
Bone Marrow Failure (Blood and lymphatic system disorders) | 0 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 29 | 40
Leukopenia (Blood and lymphatic system disorders) | 9 | 10
Neutropenia (Blood and lymphatic system disorders) | 55 | 52
Neutrophilia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 3 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 12 | 18
Acute Myocardial Infarction (Cardiac disorders) | 2 | 2
Arrhythmia (Cardiac disorders) | 0 | 1
Arteriosclerosis Coronary Artery (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 3 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 0
Cardiac Disorder (Cardiac disorders) | 0 | 1
Cardiac Failure (Cardiac disorders) | 5 | 2
Cardiac Failure Acute (Cardiac disorders) | 2 | 3
Cardiac Failure Chronic (Cardiac disorders) | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1
Cardiac Tamponade (Cardiac disorders) | 0 | 1
Cardio-Respiratory Arrest (Cardiac disorders) | 5 | 3
Cardiopulmonary Failure (Cardiac disorders) | 1 | 2
Cardiovascular Insufficiency (Cardiac disorders) | 1 | 0
Cyanosis (Cardiac disorders) | 0 | 1
Left Ventricular Dysfunction (Cardiac disorders) | 1 | 0
Left Ventricular Failure (Cardiac disorders) | 0 | 1
Myocarditis (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Pericardial Effusion (Cardiac disorders) | 0 | 1
Sinus Tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 3
Amaurosis (Eye disorders) | 1 | 0
Retinal Artery Thrombosis (Eye disorders) | 1 | 0
Vision Blurred (Eye disorders) | 0 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal Distension (Gastrointestinal disorders) | 0 | 2
Abdominal Pain (Gastrointestinal disorders) | 4 | 4
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 17 | 13
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 2
Gastrointestinal Toxicity (Gastrointestinal disorders) | 0 | 2
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Jejunal Perforation (Gastrointestinal disorders) | 0 | 1
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Mouth Ulceration (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2
Oral Pain (Gastrointestinal disorders) | 0 | 1
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 1
Peptic Ulcer (Gastrointestinal disorders) | 1 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 4 | 2
Vomiting (Gastrointestinal disorders) | 11 | 9
Abasia (General disorders) | 0 | 1
Asthenia (General disorders) | 9 | 8
Chest Discomfort (General disorders) | 0 | 1
Chest Pain (General disorders) | 2 | 1
Death (General disorders) | 1 | 7
Disease Progression (General disorders) | 0 | 1
Facial Pain (General disorders) | 1 | 0
Fatigue (General disorders) | 4 | 4
Generalised Oedema (General disorders) | 0 | 1
Malaise (General disorders) | 2 | 0
Mucosal Inflammation (General disorders) | 5 | 2
Multiple Organ Dysfunction Syndrome (General disorders) | 6 | 2
Non-Cardiac Chest Pain (General disorders) | 1 | 1
Oedema Peripheral (General disorders) | 2 | 1
Pain (General disorders) | 1 | 2
Peripheral Swelling (General disorders) | 1 | 0
Pyrexia (General disorders) | 9 | 10
Sudden Death (General disorders) | 6 | 3
Acute Hepatic Failure (Hepatobiliary disorders) | 0 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 2
Cholecystitis Chronic (Hepatobiliary disorders) | 0 | 1
Hepatic Failure (Hepatobiliary disorders) | 2 | 1
Hepatic Lesion (Hepatobiliary disorders) | 1 | 0
Hepatitis Toxic (Hepatobiliary disorders) | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 1
Hepatorenal Syndrome (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 1 | 3
Jaundice Hepatocellular (Hepatobiliary disorders) | 1 | 0
Abdominal Infection (Infections and infestations) | 0 | 1
Amoebiasis (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Biliary Sepsis (Infections and infestations) | 0 | 1
Breast Abscess (Infections and infestations) | 1 | 0
Breast Cellulitis (Infections and infestations) | 1 | 2
Bronchitis (Infections and infestations) | 0 | 1
Bronchopulmonary Aspergillosis (Infections and infestations) | 0 | 1
Candida Infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 6 | 2
Device Related Infection (Infections and infestations) | 1 | 1
Fungal Infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 3 | 0
Groin Abscess (Infections and infestations) | 0 | 1
Hepatitis Viral (Infections and infestations) | 0 | 2
Herpes Zoster (Infections and infestations) | 1 | 1
Infectious Pleural Effusion (Infections and infestations) | 0 | 1
Injection Site Abscess (Infections and infestations) | 2 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 1
Lung Infection (Infections and infestations) | 2 | 3
Mastitis (Infections and infestations) | 0 | 1
Neutropenic Infection (Infections and infestations) | 0 | 1
Neutropenic Sepsis (Infections and infestations) | 1 | 0
Oropharyngeal Candidiasis (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 0 | 2
Plasmodium Falciparum Infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 11 | 12
Pulmonary Tuberculosis (Infections and infestations) | 0 | 2
Respiratory Tract Infection (Infections and infestations) | 2 | 2
Respiratory Tract Infection Viral (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 7 | 7
Septic Shock (Infections and infestations) | 2 | 1
Tuberculosis Gastrointestinal (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 2
Viral Infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 3 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Radius Fracture (Injury, poisoning and procedural complications) | 1 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 1
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 1
Biopsy Liver (Investigations) | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 3
Dehydration (Metabolism and nutrition disorders) | 4 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 0 | 1
Electrolyte Imbalance (Metabolism and nutrition disorders) | 0 | 1
Failure to Thrive (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 4
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Soft Tissue Necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Cervix Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphangiosis Carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant Pleural Effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 10
Metastases to Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to Meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Metastases to the Respiratory System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oncologic Complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Altered State of Consciousness (Nervous system disorders) | 0 | 1
Brain Oedema (Nervous system disorders) | 0 | 1
Central Nervous System Haemorrhage (Nervous system disorders) | 1 | 0
Cerebral Haemorrhage (Nervous system disorders) | 1 | 0
Cerebral Infarction (Nervous system disorders) | 1 | 1
Cerebrovascular Accident (Nervous system disorders) | 0 | 1
Depressed Level of Consciousness (Nervous system disorders) | 2 | 3
Diabetic Hyperglycaemic Coma (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 1
Dysarthria (Nervous system disorders) | 1 | 2
Encephalopathy (Nervous system disorders) | 1 | 0
Haemorrhage Intracranial (Nervous system disorders) | 0 | 1
Haemorrhagic Cerebral Infarction (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 6 | 4
Hemiparesis (Nervous system disorders) | 1 | 1
Hemiplegia (Nervous system disorders) | 2 | 0
Hepatic Encephalopathy (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Hypoxic-Ischaemic Encephalopathy (Nervous system disorders) | 0 | 1
Iiird Nerve Paralysis (Nervous system disorders) | 1 | 0
Incoherent (Nervous system disorders) | 0 | 1
Intracranial Pressure Increased (Nervous system disorders) | 1 | 0
Ischaemic Stroke (Nervous system disorders) | 0 | 1
Loss of Consciousness (Nervous system disorders) | 1 | 1
Monoparesis (Nervous system disorders) | 0 | 1
Neuropathy Peripheral (Nervous system disorders) | 2 | 3
Paraesthesia (Nervous system disorders) | 1 | 0
Peripheral Motor Neuropathy (Nervous system disorders) | 1 | 2
Peripheral Sensorimotor Neuropathy (Nervous system disorders) | 1 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 2
Seizure (Nervous system disorders) | 6 | 4
Somnolence (Nervous system disorders) | 0 | 2
Vertebral Artery Thrombosis (Nervous system disorders) | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Device Breakage (Product Issues) | 1 | 0
Abnormal Behaviour (Psychiatric disorders) | 0 | 1
Confusional State (Psychiatric disorders) | 1 | 0
Depressed Mood (Psychiatric disorders) | 0 | 1
Mental Status Changes (Psychiatric disorders) | 2 | 0
Schizophrenia (Psychiatric disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 2 | 0
Urinary Retention (Renal and urinary disorders) | 1 | 0
Breast Mass (Reproductive system and breast disorders) | 1 | 0
Ovarian Cyst Torsion (Reproductive system and breast disorders) | 0 | 1
Pelvic Pain (Reproductive system and breast disorders) | 2 | 0
Uterine Polyp (Reproductive system and breast disorders) | 0 | 1
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Alveolitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 19
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 14 | 13
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pulmonary Artery Thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Infarction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Restrictive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis Exfoliative (Skin and subcutaneous tissue disorders) | 0 | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 1
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Stevens-Johnson Syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 2
Haemorrhage (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 2
Hypotension (Vascular disorders) | 3 | 5
Hypovolaemic Shock (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 1 | 0
Superior Vena Cava Syndrome (Vascular disorders) | 0 | 1
Vena Cava Thrombosis (Vascular disorders) | 1 | 0
Venous Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Supportive Care (SOC) (N=1045) | Epoetin Alfa (N=1051)
Anaemia (Blood and lymphatic system disorders) | 153 | 98
Leukopenia (Blood and lymphatic system disorders) | 279 | 270
Neutropenia (Blood and lymphatic system disorders) | 550 | 530
Thrombocytopenia (Blood and lymphatic system disorders) | 97 | 95
Constipation (Gastrointestinal disorders) | 40 | 53
Diarrhoea (Gastrointestinal disorders) | 189 | 180
Dry Mouth (Gastrointestinal disorders) | 46 | 57
Nausea (Gastrointestinal disorders) | 232 | 257
Stomatitis (Gastrointestinal disorders) | 79 | 71
Vomiting (Gastrointestinal disorders) | 113 | 99
Asthenia (General disorders) | 139 | 131
Fatigue (General disorders) | 215 | 201
Oedema Peripheral (General disorders) | 81 | 73
Pyrexia (General disorders) | 115 | 121
Alanine Aminotransferase Increased (Investigations) | 67 | 71
Aspartate Aminotransferase Increased (Investigations) | 66 | 77
Decreased Appetite (Metabolism and nutrition disorders) | 190 | 182
Arthralgia (Musculoskeletal and connective tissue disorders) | 81 | 56
Back Pain (Musculoskeletal and connective tissue disorders) | 54 | 55
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 59 | 66
Dysgeusia (Nervous system disorders) | 56 | 74
Headache (Nervous system disorders) | 74 | 89
Neuropathy Peripheral (Nervous system disorders) | 74 | 83
Peripheral Sensory Neuropathy (Nervous system disorders) | 111 | 97
Cough (Respiratory, thoracic and mediastinal disorders) | 95 | 122
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 74 | 77
Alopecia (Skin and subcutaneous tissue disorders) | 326 | 314

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.